CLINICAL TRIAL: NCT02103166
Title: Randomized, Masked, Placebo-controlled Clinical Trial to Evaluate the Effects of a Single Intravenous Dose of Hyoscine Bromide on the Duration and Pain in Latent and Active Labor
Brief Title: Role of Hyoscine Bromide in Latent and Active Labor
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Conditions of recruitment changed
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Montse Palacio, MD, PhD., Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 2013-001921-19
Record Dates: First submitted 2014-04-01; First posted 2014-04-03 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Labor, First Stage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyoscine bromide (Experimental): 20 mg of hyosine bromide diluted in 100 ml of physiological serum (0.9% NaCl).
  Interventions: Drug: Hyoscine bromide
- Physiological serum (Placebo Comparator): 100 ml of physiological serum (0.9% NaCl).
  Interventions: Drug: Physiological serum

INTERVENTIONS:
Drug: Hyoscine bromide — 20 mg of hyosine bromide diluted in 100 ml of physiological serum (0.9% NaCl).
  Other Names: Buscapina
  Arms: Hyoscine bromide
Drug: Physiological serum — 100 ml of physiological serum (0.9% NaCl).
  Other Names: Saline serum
  Arms: Physiological serum

SUMMARY:
The purpose of this study is to determine whether hyoscine bromide decreases the duration of the active phase of labor.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 or more.
* Term pregnancy.
* Cephalic presentation.
* Oxytocin perfusion not present at the time of inclusion.
* Uterine dynamic established.
* Abscence of high risk factors or very high risk factors for pregnancy.
* Written informed consent

Exclusion Criteria:

* Induction of labor.
* Presence of risk factors.
* Patients with hypersensitivity to the active substance or to any of the excipients or any contraindication reflected in technical report.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2014-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Time to complete dilation | One hour

CONTACTS AND LOCATIONS:
Overall Officials: Montse Palacio, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona; Mariona Rius, MD, Study Chair — Hospital Clinic of Barcelona; Ana Sandra Hernandez, MD, Study Chair — Hospital Clinic of Barcelona; Irene Teixido, MD, Study Chair — Hospital Clinic of Barcelona; Irene Vives, MD, Study Chair — Hospital Clinic of Barcelona; Midwives Collaborative Group HCP, Study Chair — Hospital Clínic
Locations (1):
- Hospital Clínic, Barcelona, Barcelona, Spain